CLINICAL TRIAL: NCT00673140
Title: Phase 1 Study to Determine the Efficacy of Using Far Infrared Radiation for the Control, Management and Treatment of Amyotrophic Lateral Sclerosis (ALS) or Lou Gehrig's Disease
Brief Title: Far Infrared Irradiation for Control, Management and Treatment of Amyotrophic Lateral Sclerosis (ALS)
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: GAAD Medical Research Institute Inc. (Other)
Responsible Party: Dr. Kwasi Donyina/Founder and President, GAAD Medical Research Institute Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GAAD-ALS-CTP1
Record Dates: First submitted 2008-05-06; First posted 2008-05-07 (Estimated); Last update posted 2009-08-17 (Estimated); Status verified 2009-08

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: ALS (Amyotrophic Lateral Sclerosis); Amyotrophic Lateral Sclerosis With Dementia; Amyotrophic Lateral Sclerosis, Guam Form; Dementia With Amyotrophic Lateral Sclerosis; Gehrig's Disease; Guam Form of Amyotrophic Lateral Sclerosis; Lou Gehrig Disease
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Radiation: Far Infrared Radiation (5μm to 20μm wavelength)
  Interventions: Radiation: Far Infrared Radiation (5μm to 20μm wavelength); Radiation: Far infrared radiation

INTERVENTIONS:
Radiation: Far Infrared Radiation (5μm to 20μm wavelength) — Radiation: Far Infrared Radiation (5μm to 20μm wavelength). Far Infrared radiation for 30 to 40 minutes per treatment session.
  Other Names: Radiation: Far Infrared Radiation (5μm to 20μm wavelength)
Radiation: Far infrared radiation — Far infrared radiation at a frequency of 5 microns to 20 microns for 30 to 40 minutes per session.

SUMMARY:
Amyotrophic Lateral Sclerosis (ALS, sometimes called Lou Gehrig's s Disease, or Maladie de Charcot) is a progressive, usually fatal, neurodegenerative disease caused by the degeneration of motor neurons, the nerve cells in the central nervous system that control voluntary muscle movement.

This study will investigate the use of far infrared radiation for the control, management and treatment of ALS.

DETAILED DESCRIPTION:
As a motor neuron disease, ALS causes muscle weakness and atrophy throughout the body as both the upper and lower motor neurons degenerate, ceasing to send messages to muscles. Unable to function, the muscles gradually weaken, develop fasciculations (twitches) because of denervation, and eventually atrophy due to that denervation. The patient may ultimately lose the ability to initiate and control all voluntary movement except of the eyes.

Observations from our research studies indicate that, far infrared rays provide energy to the body, improve the autonomic functions of the nervous system, restore the functions of the endocrine system, strengthen the immune system, improve blood circulation and increase the level of oxygen in the cells and promote the regeneration of muscle cells, nerves and brain cells.

It is hereby postulated that irradiation using far infrared, with wavelength between 5 to 20 microns, of the central nervous system, the endocrine system and the whole body could prevent, control, manage or possibly lead to complete rehabilitation of people who have ALS.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ALS

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2008-05; Primary Completion 2010-05 (Estimated); Study Completion 2010-06 (Estimated)

PRIMARY OUTCOMES:
Therapy for ALS | 2 years

SECONDARY OUTCOMES:
Rehabilitation of ALS patients | 2 Years

CONTACTS AND LOCATIONS:
Overall Officials: Ken Nedd, M.D., Principal Investigator — GAAD Medical Research Institute Inc.
Locations (1):
- The Centre for Incurable Diseases, Toronto, Ontario, Canada